CLINICAL TRIAL: NCT06152055
Title: Clinicopathological Profile of Head and Neck Cancers in Army Hospital of Nepal - A Retrospective Study
Brief Title: Clinicopathological Profile of Head and Neck Cancers in Army Hospital of Nepal
Status: Completed | Type: Observational
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Anupama Marasini, Intern Doctor, Tribhuvan University, Nepal
Other Study IDs: 245
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a observational study conducted at the department of Ear ,Nose and Throat -Head and Neck Surgery (ENT-HNS) of Shree Birendra Hospital ,a tertiary health care centre of Nepal. Head and Neck cancers are the sixth most common cancer in the world. Data was collected from the medical records of Head and Neck Cancer patients who underwent treatment between May 2022 to April 2023.The main aim of the study was to know about the common cancers of head and neck region and their distribution according to the site. Also to know the stage of the presentation with treatment modalities in the tertiary health care centre of Nepal.

DETAILED DESCRIPTION:
This is a retrospective study to know the prevalence of Head and Neck Cancer at the department of ENT- Head and Neck Surgery of Shree Birendra Hospital ,a tertiary health care centre of Nepal .Head and neck cancers are malignant neoplasms that develops in oral cavity, nasal cavities, paranasal sinuses,nasopharynx, oropharynx, hypopharynx, ear, scalp, salivary gland and neck,Data was collected from the medical records of Head and Neck Cancer patients who underwent treatment between May 2022 to April 2023. Data considered of demographic details of age, sex, diagnosis, subsite specific Head and Neck Cancers, treatment modality and histopathology. The data was analyzed using Stastical Package for Social Sciences (SPSS) version 22. Pearson's chi-square test was applied and p value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All histologically proven cases of head and neck region.

Exclusion Criteria:

* Patient's record with incomplete data.

Ages: 17 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population was selected from the tertiary care centre of Nepal.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Age - wise Distribution of Head and Neck Cancers (HNCs) | 1 year
  Age - wise Distribution of Head and Neck Cancer
: Distribution of HNCs according to subsite | 1 year
  Distribution of Head and Neck Cancers according to the subsite
Histopathology of HNCs | 1 year
  Histopathology of Head and Neck Cancer
Tumor, Nodes, Metastasis (TNM) staging of HNC | 1 year
  Staging at presentation of Head and Neck Cancer
Treatment provided to HNC patients | 1 year
  Treatment Modalities of Head and Neck Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Reeba Karki, MS, Principal Investigator — Shree Birendra Hospital
Locations (1):
- Shree Birendra Hospital, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data to protect the privacy of the participants.

REFERENCES:
- [Background] Chin D, Boyle GM, Porceddu S, Theile DR, Parsons PG, Coman WB. Head and neck cancer: past, present and future. Expert Rev Anticancer Ther. 2006 Jul;6(7):1111-8. doi: 10.1586/14737140.6.7.1111. PMID 16831082